CLINICAL TRIAL: NCT06906757
Title: Preterm Rupture of Membranes Optimising Antibiotics Trial (PROMOAT). A Pregnancy Domain Within PLATIPUS.
Brief Title: Preterm Rupture of Membranes Optimising Antibiotics Trial
Acronym: PROMOAT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Melbourne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: P-P01-PROMOAT
Record Dates: First submitted 2025-02-18; First posted 2025-04-02 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-02

CONDITIONS: PPROM; Preterm
Keywords: Pregnancy, Preterm, PPROM, Antibiotics; chorioamnionitis
MeSH Terms: conditions — Preterm Premature Rupture of the Membranes; Premature Birth; Chorioamnionitis | interventions — Erythromycin; Azithromycin; Amoxicillin

STUDY DESIGN:
Intervention Model Description: PROMOAT is a domain within the PLATIPUS adaptive platform trial (NCT06461429).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All parties will be blinded to the assigned intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Erythromycin 250mg + placebo (Active Comparator): Erythromycin 250mg, four times a day, for 7 days. Oral preparation only.
  Placebo tablets instead of penicillin for blinding purposes.
  Interventions: Drug: Erythromycin 250mg + placebo
- Azithromycin 500mg + placebo (Active Comparator): Azithromycin 500mg daily for 7 days. Oral preparation only.
  Placebo tablets instead of penicillin for blinding purposes.
  Interventions: Drug: Azithromycin 500mg + placebo
- Erythromycin 250mg and Amoxicillin 500mg (Active Comparator): Erythromycin 250mg, four times a day AND Amoxicillin 500mg three times a day, for 7 days. Oral preparations only.
  Interventions: Drug: Erythromycin 250mg and Amoxicillin 500mg

INTERVENTIONS:
Drug: Erythromycin 250mg + placebo — Antibiotic.
  Arms: Erythromycin 250mg + placebo
Drug: Azithromycin 500mg + placebo — Antibiotic.
  Arms: Azithromycin 500mg + placebo
Drug: Erythromycin 250mg and Amoxicillin 500mg — Antibiotics.
  Arms: Erythromycin 250mg and Amoxicillin 500mg

SUMMARY:
The goal of this clinical trial is to learn which antibiotic regimen works best to prevent infection in pregnant women whose waters break early (preterm, pre-labour rupture of membranes, or PPROM) and assess the health outcomes of babies born to pregnant women who have received these antibiotics.

PROMOAT aims to answer the question: Which antibiotic or combined antibiotic regimen most effectively prevents infection in pregnant women with PPROM < 37+0 weeks' gestation.

Researchers will compare three antibiotic regimens already used in clinical practice to prevent infection in pregnant women with PPROM.

Participants will be randomly allocated to the antibiotic regimen they will follow for seven days, or until birth (whichever is earlier). All antibiotics will be taken orally.

Neonatal health outcomes will be collected at 42 weeks postmenstrual age and maternal birth and postpartum care outcomes assessed at 42 days postpartum.

Questionnaires will capture maternal mood at time of consent and at 42 days postpartum. Antibiotic tolerance will be assessed at the time antibiotic treatment is ceased.

This trial will be undertaken as part of the PLATIPUS trial (NCT06461429).

DETAILED DESCRIPTION:
PROMOAT aims to determine which of the most common antibiotic regimens are most effective in preventing infection in pregnant people with PPROM to improve health outcomes for their infants. PROMOAT is a pregnancy domain within the PLATIPUS adaptive platform trial (NCT06461429).

Preterm prelabour rupture of membranes (PPROM) precedes 30-40% of spontaneous preterm births and is an important cause of maternal and neonatal infection. Membrane rupture provides an entry point for microbes from the vagina to ascend into the uterine cavity, exposing the mother and the fetus to infectious pathogens leading to poor maternal and neonatal outcomes. Mothers with PPROM are at increased risk of haemorrhage, hysterectomy, sepsis, intensive care admission and death. Preterm infants exposed to in-utero infection are at higher risk of poor short- and long-term outcomes, including neonatal sepsis, neurodevelopmental delay, cerebral palsy, chronic lung disease and death.

Neonatal sepsis is the third most common cause of newborn deaths (~340,000 per year) and prevention is a major research priority, Neonatal sepsis due to pathogens acquired after PPROM may present in the first days of life and result in bacteraemia, pneumonia and meningitis. The most common pathogens associated with early-onset neonatal sepsis are Streptococcus agalactiae (aka Group B Streptococcus: GBS), Escherichia coli and Ureaplasma sp. Mortality is highest in the most immature infants, with a 54% case fatality rate in infants born before 24 weeks' gestation.

The goal in managing pregnancies complicated by PPROM is to prolong the pregnancy to enable fetal maturity without an increased risk of infection (acquired while the fetus remains in utero). Antibiotic prophylaxis has been shown to increase latency to birth but there is limited evidence to guide antibiotic choice to prevent infection in PPROM.

In PROMOAT, pregnant women with PPROM will be randomly assigned to receive one of the three intervention arms:

* Erythromycin
* Azithromycin, or
* Erythromycin and Amoxicillin.

Health outcomes will be assessed using the PLATIPUS Ordinal Outcome Scale, at 42 weeks' postmenstrual age or discharge home, whichever is earliest.

A short questionnaire at Day 7 (or birth, whichever is earlier) will measure compliance and antibiotic tolerance. A maternal and family health questionnaire will be collected at Day 42 postpartum.

ELIGIBILITY:
PLATFORM ELIGIBILITY

Participants must meet all core PLATIPUS platform inclusion criteria:

* Considered to be at risk of birth before 37 weeks gestation (spontaneous and provider-initiated)
* Receiving pregnancy care at a participating site (hospital) at the time of eligibility assessment and
* Meet eligibility criteria for one or more platform domains.

Participants will be excluded from participation if they meet any core PLATIPUS platform exclusion criteria:

* Inability to consent for themselves
* Perinatal death is deemed to be imminent and inevitable during the next 24 hours (at time of screening).

Pregnant women and people who meet ALL of the core platform inclusion criteria and none of the exclusion criteria will be considered for PROMOAT-specific eligibility.

PROMOAT-SPECIFIC ELIGIBILITY

Platform-eligible participants must meet all PROMOAT-specific inclusion criteria:

1. Women with singleton or multiple pregnancies complicated by preterm prelabour rupture of membranes (PPROM) < 37+0 weeks' gestation as determined by the treating clinician and standard criteria:

   * Maternal history consistent with loss of fluid per vagina
   * Evidence of a pool of fluid in the vagina on sterile speculum examination
   * +/- positive testing for IGFBP-1 (Actim PROM) or PAMG-1 (Amnisure) AND
2. Are eligible for at least two treatment arms within the domain
3. The fetus/fetuses are alive at randomisation
4. The pregnancy is continuing and active neonatal management is planned.

Participants will be excluded from participation if they meet core PLATIPUS platform exclusion criteria:

* Inability to consent for themselves OR
* Perinatal death is deemed to be imminent and inevitable during the next 24 hours (at time of screening).

Participants will be excluded from participation if they meet any PROMOAT-specific exclusion criteria:

1. Antibiotic treatment for > 24 hours administered with the aim of preventing infection from PPROM
2. Suspected maternal or fetal infection (chorioamnionitis)
3. Maternal or fetal indication for immediate birth
4. Established preterm labour (cervical dilatation ≥ 3cm AND regular contractions)
5. No appropriate antibiotic available within domain intervention arms due to allergy, contraindications, drug interactions, drug availability, or previous history of antibiotic-resistant infection/s
6. Women with a previous infant affected by GBS sepsis
7. Major congenital fetal anomaly.

Platform-eligible participants who meet all PROMOAT-specific inclusion criteria and none of the PROMOAT-specific exclusion criteria will be eligible to participate in PROMOAT.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3900 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2029-12 (Estimated); Study Completion 2050-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants who progress by at least one level higher on the PLATIPUS Ordinal Outcome Scale [PLATIPUS Core Primary Outcome] | At any time prior to 42 weeks' postmenstrual age or first discharge home from hospital (whichever is earlier).]
  The PLATIPUS-Ordinal Outcome Scale ranks the most severe core short-term infant health outcome in the specified time frame.
  Levels 1-15: 1= Well, liveborn infant; 2= Neonatal unit admission for <48 hours; 3= Neonatal unit admission for >/= 48 hours; 4= Non-invasive respiratory support or oxygen therapy for ≥ 4 hours & < 5 days; 5= Non-invasive respiratory support or oxygen therapy >/= 5 days; 6= Mechanical ventilation via endotracheal tube for ≥ 4 hours & <7 days; 7= Mechanical ventilation via endotracheal tube for >/=7 days; 8= Moderate respiratory morbidity; 9=Necrotising enterocolitis AND/OR Sepsis; 10= Severe Respiratory Morbidity; 11= Major Surgery; 12= Brain Injury; 13= TWO of severe respiratory morbidity OR major surgery OR brain injury; 14= Severe respiratory morbidity & major surgery & brain injury; 15 = Death.

SECONDARY OUTCOMES:
Time (randomisation) to birth | From randomisation to birth
  Number of days from randomisation to birth.
Estimated antepartum/intrapartum/postpartum (< 24 hours) blood loss | Less than 24 hours of birth.
  Estimated antepartum/intrapartum/postpartum (<24 hours of birth) blood loss.
Rate of clinical chorioamnionitis | To birth.
  Clinical chorioamnionitis Clinical suspicion of intra-amniotic infection such as: maternal fever (>/= 38C AND 2 of maternal tachycardia (> 100 beats/min), fetal tachycardia 26,27(> 160 beats/min), uterine tenderness, purulent/malodorous amniotic fluid, maternal leukocytosis (white blood cell count >/= 15,000/mm3) AND Antibiotics commenced for treatment for clinically suspected chorioamnionitis.
Rate of histological chorioamnionitis/funisitis | To birth
  Histological chorioamnionitis/funisitis
  • Presence of inflammation in the placenta, chorion, umbilical cord and/or amnion with or without fetal inflammatory response defined according to staging of maternal (MIR) or fetal inflammatory response (FIR).
Rate of puerperal infection | From birth to day 42 postpartum
  Puerperal infection Infection of the maternal genital tract, urinary tract and wound infection from birth to day 42 postpartum AND Antibiotic treatment commenced
Rate of early onset neonatal sepsis | Within 48 hours of birth.
  Isolation of a bacterial or fungal organism from at least one of blood or CSF culture or by PCR sampled within 48 hours of birth AND after consideration of clinical and laboratory evidence, a decision is made to give the infant antibiotics with therapeutic intent against this organism for >5 days
Duration of neonatal antibiotic use commenced within 48 hours of birth. | Within 48 hours of birth.
  Duration of neonatal antibiotic treatment commenced within 48 hours of birth.
Number of days of maternal antibiotic prescription after birth to day 42 postpartum | From birth to Day 42 postpartum
  Estimated cumulative days of maternal antibiotic use from birth to day 42 postpartum

OTHER OUTCOMES:
Core Secondary Outcome 1: Number of maternal deaths within 42 days postpartum | From birth to 42 days postpartum
  Number of mother (or birth parent) deaths within 42 days of birth.
Core Secondary Outcome 2: Rate of severe maternal morbidity | From platform entry to 42 days postpartum
  Maternal or pregnant person morbidity is defined as: unplanned ICU admission, sepsis, eclampsia, amniotic fluid embolism, pregnancy-related hysterectomy, severe primary postpartum haemorrhage, uterine rupture, cardiac arrest, mechanical ventilation (not for birth), stroke.
Core Secondary Outcome 3: Duration of hospitalisation | From date of platform entry to date of first discharge home from hospital (birth admission).
  Duration of maternal or pregnant person hospitalisation, in days, after platform entry
Core Secondary Outcome 4: Rate of readmission to hospital | From first discharge home from hospital (birth admission) to 42 days postpartum.
  Rate of readmission to hospital, after first discharge home from hospital, within 42 days postpartum.
Core Secondary Outcome 5: Rate of mode of birth | At birth
  Rates of vaginal birth vs assisted vaginal birth vs caesarean birth.
Core Secondary Outcome 6: Infant gestational age at birth. | From estimated date of delivery to date of birth.
  Calculated infant gestation age based on estimated date of delivery and date of birth.
Core Secondary Outcome 7: Infant birth weight z-score. | At birth
  Z-score generated from infant weight at birth and gestational age at birth.

CONTACTS AND LOCATIONS:
Overall Officials: Clare Whitehead, MBChB, PhD, Principal Investigator — University of Melbourne and Royal Women's Hospital (Melbourne)

IPD SHARING:
Plan to Share IPD: Yes
Data sharing will align with PLATIPUS (NCT06461429) policy. Version 1, Apr-2024
  Once data unblinding no longer compromises the integrity of the trial, a de-identified data set collected for the analysis of domains within PLATIPUS will be made available.
  Conditions
  1. All domains in which the participant is co-enrolled are closed to recruitment* (*Where one or more domains in which a participant is co-enrolled are not yet closed to recruitment, the participant's data may be provided, without the treatment code, to prevent unblinding in unfinished domains).
  2. Primary domain conclusions/analyses have been published, AND
  3. The 2-year follow-up of participants within the domain/s of interest is/are complete.
  Supporting materials (Core Protocol, Domain-Specific Appendices, Data Dictionaries and Domain-Specific Statistical Analysis Plans) will be available.
  Contact: University of Melbourne - info@platipustrial.org.
Supporting Information: Study Protocol, SAP
Time Frame: This is estimated to be approximately six months following the completion of the two-year follow-up of domain participants.
Access Criteria: To be determined. Access requests will be subject to review by trial subcommittees. The Trial Steering Committee will approve or disapprove requests. A Data Transfer Agreement and Authorship Agreement signed by relevant parties and evidence of ethical approval will be required.